CLINICAL TRIAL: NCT03357601
Title: The Effect of High Intensity Interval vs Moderate Continuous Endurance Exercise Training on Program Adherence
Brief Title: High Intensity Interval Training vs Moderate Continuous Endurance Exercise Training on Program Adherence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Professor, Western University, Canada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110476
Record Dates: First submitted 2017-11-17; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Physical Activity; Fat Burn
Keywords: High Intensity Interval; Moderate Endurance Exercise; Fat Loss; Endurance Capacity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Each participant will be match-paired to either HIIT or MCEET group based on their time to complete a mile run. There will be rank from 1 to 40, where number one will be assigned randomly to one group while two goes to the other group. Then, number three goes to the second group and fourth is assigned to the first group. Alternating patterns will be continued thereafter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (Experimental): six 20 second bouts of high intensity interval exercise (HIIT) separated by 2 minutes of active recovery with 3 minutes and warm up and cool down on the treadmill, three times per week for five weeks
  Interventions: Behavioral: HIIT
- MCEET (Experimental): 14 minutes of Moderate Endurance Training with 3 minutes and warm up and cool down on the treadmill, three times per week for five weeks
  Interventions: Behavioral: MCEET

INTERVENTIONS:
Behavioral: HIIT — The participant will perform HIIT where they will warm up for 3 minutes at 30% maximum heart rate (MHR), followed by 20 seconds of high intensity interval exercise at an all out intensity separated by 2 minutes of active recovery at 30% MHR. The interval will be repeated six times. Once completing all six intervals, participants will cool down for 3 minutes. This training program will be performed three times per week for five weeks.
  Arms: High Intensity Interval Training
Behavioral: MCEET — The participant will perform MCEET, where they will warm up for 3 minutes at 30% maximum heart rate (MHR), followed by 14 minutes of moderate, continuous endurance exercise at 70% MHR. Participants will cool down for 3 minutes. This training program will be performed three times per week for five weeks.
  Arms: MCEET

SUMMARY:
This study examines whether high intensity interval training (HIIT) or moderate, continuous endurance exercise training (MCEET) results in greater program adherence when matched for session time. Body composition and endurance capacity will also be measured to identify any significant changes among two exercise groups. It is hypothesized that HIIT will result in greater program adherence as well as greater improvements in body composition and endurance capacity. Both exercise groups will complete 20 minutes sessions (which include exercise) three times per week for five week. The first week will be supervised by study investigators while the remainder of the study will be unsupervised in order to examine how free-living individuals adhere to two exercise programs. There will be no attempt to restrict food intake during the exercise intervention. Body composition will be measured by densitometry [body mass/body volume] using a BodPod. Endurance capacity will be assessed using a mile run. Two validated questionnaires [Physical activity enjoyment scale and Exercise adherence ratings scale] as well as heart rate data (recorded before, during and after each training sessions) will be used to confirm exercise adherence. These data may help us determine the optimal type of exercise program to maintain healthy body composition.

DETAILED DESCRIPTION:
Upon completing informed consent, all the eligible participants will have their body composition measured at the Exercise Nutrition Research Laboratory, Western University, using non-invasive air displacement plethysmography (BodPod). This requires participants to sit in a chamber while space [volume] their bodies take up is assessed. This along with their body mass allows body density [d=m/v] and body composition to be determined pre and post the 5-week exercise intervention. Upon completing the body composition measurements, participants will have their endurance capacity assessed by performing a timed one-mile run (which will be used as an index of their endurance capacity). Participants will be advised to dress appropriately for physical activity including proper footwear.

Each participant will be matched to either HIIT or MCEET group based on their one-mile run time. The HIIT group will perform six, 20-second bouts of high-intensity interval exercise separated by 2 minutes of active recovery (walking) while the MCEET group will perform 14 minutes of continuous endurance exercise at 70% of Maximum Heart Rate (MHR). Both exercise protocols will include 3 minutes of warm up and cool down at a 30% MHR, for a total of 20 minutes for each treatment. The first week of the exercise intervention will consist of one-on-one supervised treadmill training, three times per week in the lab. From week two to five, participants will follow the same exercise program on their own at their preferred gym three times per week in order to examine free-living individuals adhere to two exercise programs.

All participants will log their heart rate before, during, and immediately after each training session using a free heart rate monitor mobile App to ensure safety and achievement of their targeted heart rate. Further, they will complete two validated questionnaires [physical activity enjoyment scale and exercise adherence rating scale] as well ratings of perceived exertion scale after the 6th, 9th and 15th session. Finally, no attempt will be made to modify the participants daily diet, but a 3-day food log will be collected to assess food intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 19-35 years old
* Engage in physical activity less than three times per week
* Must have access to the gym
* Must have smartphones (such as Android, Cat phone, Google Nexus, Samsung Galaxy, iPhone, Microsoft Lumia, myTouch or Phablets)
* Must have access to Apps (such as MyFitnessPal, Rise Up, Calorific, My Diet Coach, Yazio, On The Regimen, See How You Eat, Lost It, MyNetDiary or MyPlate)
* Must be able to run a mile

Exclusion Criteria:

* Diabetic
* Pregnant
* History of fainting
* Low and high blood pressure
* Heart disease
* Migraines
* Experience with heartburn
* Smokers
* Respiratory diseases
* Engage in physical activity more than two times per week
* Answering YES to any questions from page 1 of GAQ

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-03 (Estimated); Primary Completion 2018-02-07 (Estimated); Study Completion 2018-02-14 (Estimated)

PRIMARY OUTCOMES:
Program Adherence | 5 weeks
  Physical Activity Enjoyment Scale assess levels of exercise enjoyment based on 18 questions on a 1 to 7 Likert Scale
Program Adherence | 5 weeks
  Exercise Adherence Rating Scale measures adherence to prescribed exercise program based on 6 questions on a 0 to 4 Likert Scale

SECONDARY OUTCOMES:
Body Composition | 5 weeks
  A whole body densitometry (BodPod) measures body mass, fat mass and non-fat mass to determine body density which then gives body composition
Endurance Capacity | 5 weeks
  A mile run performance is an indication for a relative VO2 max.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western University, Canada
Locations (1):
- 3M Centre, Room 2225, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillen JB, Martin BJ, MacInnis MJ, Skelly LE, Tarnopolsky MA, Gibala MJ. Twelve Weeks of Sprint Interval Training Improves Indices of Cardiometabolic Health Similar to Traditional Endurance Training despite a Five-Fold Lower Exercise Volume and Time Commitment. PLoS One. 2016 Apr 26;11(4):e0154075. doi: 10.1371/journal.pone.0154075. eCollection 2016. PMID 27115137
- [Background] Macpherson RE, Hazell TJ, Olver TD, Paterson DH, Lemon PW. Run sprint interval training improves aerobic performance but not maximal cardiac output. Med Sci Sports Exerc. 2011 Jan;43(1):115-22. doi: 10.1249/MSS.0b013e3181e5eacd. PMID 20473222
- [Background] Thum JS, Parsons G, Whittle T, Astorino TA. High-Intensity Interval Training Elicits Higher Enjoyment than Moderate Intensity Continuous Exercise. PLoS One. 2017 Jan 11;12(1):e0166299. doi: 10.1371/journal.pone.0166299. eCollection 2017. PMID 28076352
- See also: Three Minutes of All-Out Intermittent Exercise per Week Increases Skeletal Muscle Oxidative Capacity and Improves Cardiometabolic Health — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0111489
- See also: Sample size calculation — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2876926/
- See also: Attrition and Adherence Rates of Sustained vs. Intermittent Exercise Interventions — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3181282/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT03357601/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT03357601/ICF_001.pdf